CLINICAL TRIAL: NCT07205939
Title: Remote Assessment of the Permanent Site After Cesarean Section: A Randomized Controlled Trial
Brief Title: Evaluation of Surgical Site Infection After Cesarean Section
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sibel Bulut Haklı (Other)
Responsible Party: Sponsor-Investigator, Sibel Bulut Haklı, PhD Candidate, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ISU-CS-23-277
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Surgical Infection; Cesarean Section Wound
Keywords: mobile application; cesarean section; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Usual Care) - routine postpartum wound care instructions and scheduled follow-up. (No Intervention)
- Mobile App Telemonitoring + Standard Care (Experimental)
  Interventions: Device: Mobile Application usage

INTERVENTIONS:
Device: Mobile Application usage — Articipants complete a brief symptom questionnaire and upload a standardized photo of the cesarean incision on postpartum days 3, 7, and 15 (±1 day) via the study mobile platform. Patients will be reminded remotely on these mandatory days. They will be informed that if they have concerns about the wound outside of these mandatory days, they can use the app and share their survey and image data.
  The surveys and images uploaded to the app will be evaluated by the researcher and reviewed by a clinician. Retakes will be requested for photos that are not of sufficient quality for evaluation. Clinical recommendations after review will be based on the patient's reported symptoms, and the wound images will provide additional information on this topic. One month after the cesarean section, all participants will be contacted by the researcher. They will be asked about the current status of their wounds and a patient satisfaction survey will be administered.
  Other Names: SurgiMomma
  Arms: Mobile App Telemonitoring + Standard Care

SUMMARY:
This study aims to investigate surgical site monitoring after cesarean section using a mobile application currently being developed. This mobile application aims to facilitate early diagnosis of surgical site infection, reduce clinic visits for wound monitoring, and consequently reduce labor, travel, and care costs. In this context, a randomized controlled design will be conducted between the study and control groups to compare surgical site infection rates, time to diagnosis, number of clinic visits, frequency of hospitalization, care costs, and patient satisfaction.

DETAILED DESCRIPTION:
While birth occurs spontaneously and naturally at the end of pregnancy due to a woman's normal physiology, intervention is required if a condition endangers the pregnant woman or the fetus. Cesarean section is the surgical procedure of choice when vaginal birth threatens maternal or fetal health, or when vaginal birth is not possible for various reasons. Cesarean section rates (both emergency and elective) range from 5% to 20%, and rates continue to increase in all countries. The frequency of Cesarean sections has increased by 75% over the last 15 years. The term surgical site infection (SSI) was coined by the Surgical Wound Infection Task Force in 1992. In its broader sense, SSI is classified as an infection that occurs within 30 days after surgery, either due to an incision or deep tissue injury. Bacteria entering through the incision line during surgery are the cause of the spread of potentially life-threatening surgical site viruses each year and contribute to the rise in antibiotic resistance. In low- and middle-income families, 11% of patients undergoing surgery develop this condition during this time.

More than 2 million laparotomies are performed annually for benign conditions in the United States. More than half of these (1 million cesarean sections and 500,000 hysterectomies) are obstetric and gynecological procedures. Although precise figures for similar data are not available in Turkey, it is known that the frequency of cesarean sections is quite high. Among all OECD (Organization for Economic Cooperation and Development) countries, Turkey has the second-highest cesarean section rate at 57.3%. The estimated incidence of SSI ranges from 3% to 15% for cesarean sections and 3% to 8% for abdominal hysterectomies. 3% to 14% of cesarean sections are complicated by wound seroma and hematoma. In Africa, up to 20% of cesarean section patients develop a wound infection, compromising their health and their ability to care for their babies. Post-cesarean SSI can be associated with many factors. These include age, body mass index (BMI), inadequate antenatal care, smoking, diabetes mellitus, hypertensive disorders, and multiple pregnancies, as well as intrapartum risk factors such as emergency cesarean section, prolonged labor, premature rupture of membranes, frequent vaginal examinations, and chorioamnionitis. Western sources estimate hospital expenses per wound. Therefore, the direct costs of laparotomy wounds in obstetrics and gynecology can reach $180 to $500 million annually. These figures do not include home wound care and nursing, dressings, additional office visits, lost work, and physical and psychosocial costs for the patient. In the short term, wound dehiscence prolongs postoperative pain and healing time, while also contributing to protein and nitrogen loss. In the long term, a severed, infected wound can lead to scarring and an increased risk of herniation. The emotional and social consequences are less well known, and the impact on the development of chronic pain is unknown. Telehealth is the sharing of health data, care information, and education between healthcare personnel and patients, students, and other healthcare professionals via telecommunications, using telephones, computers, interactive television, or a combination of these. The COVID-19 pandemic, in particular, has highlighted the need for the creation and expansion of telehealth systems. Telehealth systems aim to identify changes in patients' vital signs early, provide early intervention, reduce the number of home visits, reduce the number of emergency room and outpatient clinic visits, reduce hospitalization rates, hospitalization duration, and care costs, while also improving patient self-care. This study aimed to investigate surgical site control after cesarean section using a mobile application being developed.

ELIGIBILITY:
Inclusion Criteria: Women who have had a Caesarean section Owning a smartphone with internet access Ages 18-45 Providing informed consent Adequate Turkish reading comprehension

Exclusion Criteria: Presence of illnesses that prevent the use of the online survey/application (visual impairment, neuropsychiatric illnesses, etc.).

Failure to comply with working conditions (not completing forms, missing forms, etc.)

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) within 30 days (CDC criteria) | 30 days post-cesarean
  SSI status adjudicated per CDC criteria by a blinded outcomes assessor.

CONTACTS AND LOCATIONS:
Overall Officials: SİBEL BULUT HAKLI, Principal Investigator — Istinye University
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
e are evaluating the feasibility of sharing a de-identified individual participant dataset excluding raw wound photographs, pending final ethics approval and explicit consent language. If feasible, the dataset would include group assignment, baseline characteristics, primary and secondary outcomes, and derived image variables (e.g., erythema/drainage present vs absent). Direct identifiers will be removed, dates will be shifted, and rare categories top-coded. This record will be updated prior to publication of the primary results.

REFERENCES:
- [Background] Rochon M, Jawarchan A, Fagan F, Otter JA, Tanner J. Image-based digital post-discharge surveillance in England: measuring patient enrolment, engagement, clinician response times, surgical site infection, and carbon footprint. J Hosp Infect. 2023 Mar;133:15-22. doi: 10.1016/j.jhin.2023.01.001. Epub 2023 Jan 13. PMID 36642336
- [Background] McLean KA, Sgro A, Brown LR, Buijs LF, Daines L, Potter MA, Bouamrane MM, Harrison EM. Evaluation of remote digital postoperative wound monitoring in routine surgical practice. NPJ Digit Med. 2023 May 5;6(1):85. doi: 10.1038/s41746-023-00824-9. PMID 37147462
- [Background] McLean KA, Mountain KE, Shaw CA, Drake TM, Pius R, Knight SR, Fairfield CJ, Sgro A, Bouamrane M, Cambridge WA, Lyons M, Riad A, Skipworth RJE, Wigmore SJ, Potter MA, Harrison EM; TWIST Collaborators. Remote diagnosis of surgical-site infection using a mobile digital intervention: a randomised controlled trial in emergency surgery patients. NPJ Digit Med. 2021 Nov 18;4(1):160. doi: 10.1038/s41746-021-00526-0. PMID 34795398